CLINICAL TRIAL: NCT01816490
Title: A Phase II, Multi-center, Open-label, Interventional Study to Evaluate the Safety of Intravenous Silibinin (iSIL) and Its Effect on the Hepatitis C Virus Load in Treatment-experienced HCV-HIV Co-infected Individuals With Advanced Liver Fibrosis in the Swiss HIV Cohort Study (SHCS)
Brief Title: THISTLE - The HIV-HCV Silibinin Trial
Acronym: THISTLE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: THISTLE
Record Dates: First submitted 2013-03-08; First posted 2013-03-22 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2013-09

CONDITIONS: HIV; Hepatitis C
MeSH Terms: conditions — Hepatitis C

INTERVENTIONS:
Drug: Intravenous Silibinin (iSIL)

SUMMARY:
Chronic hepatitis C virus (HCV) is a major cause of morbidity and mortality worldwide with an estimated number of 180 million infected patients. Until 2012 the current standard of care (SOC) treatment of patients with chronic hepatitis C was a 24 to 72 weeks therapy with pegylated interferon- and ribavirin (PR). In 2012, the protease-inhibitors (PI's) telaprevir and boceprevir as first directly acting HCV drugs have been approved by the local Swiss authority for hepatitis C mono-infected and HCV-HIV-co-infected individuals. However, therapy success is strongly limited in null-responders (NR) to previous PR. Treatment of HCV-HIV co-infected individuals with the new PI's is accompanied by additional challenges (e.g. drug-drug interactions, toxicity, high pill burden). Patients with advanced fibrosis are at highest risk for decompensated liver disease and hepatocellular carcinoma (HCC) and prompt initiation of treatment is strongly recommended. Recently, data in mono-infected patients showed, that in prior non responders a 12 week course of a triple therapy (TT) with telaprevir and PR followed by another 24 weeks of PR resulted in an sustained virologic response (SVR) of only 29%. In HCV-HIV co-infected non-responders with unfavourable preconditions (e.g. HCV-genotype 1, interleukin 28 B non-CC genotype, advanced liver fibrosis, high baseline HCV viral load) SVR after TT is even expected to be lower. These patients urgently need additional therapeutic options with the goal to eradicate HCV in order to prevent further fibrosis progression and to reduce morbidity and mortality. A promising substance in the field of drugs targeting the HCV replication is silibinin. Silibinin is the main component of silymarin, an extract of the milk thistle Silybum marianum. Intravenous silibinin (iSIL) targets multiple steps in the virus life cycle and exhibits anti-oxidant, anti-inflammatory, anti-viral and immunomodulatory properties. iSIL inhibits the HCV NS5B polymerase activity directly or by interfering with the binding of RNA to this enzyme. In addition, iSIL appears to block virus entry, virus transmission and virus secretion.In 2008 Ferenci et al. for the first time reported the substantial clinical antiviral-effect of intravenous silibinin (iSIL) against HCV in PR non-responders. The administration of 20mg/kg iSIL in 20 patients led to a highly significant decrease in viral load. We intend to investigate the effect and tolerability of iSIL in HIV-HCV co-infected individuals with advanced liver fibrosis and previous non- or partial response to SOC. All included study-subjects will receive a lead-in therapy with iSIL in a dosage of 20mg/kg/day (expressed as silibinin concentration) once a day for 14 days. At the end of the THISTLE study, i.e. after the day of completion of the 14-day iSIL administration (day 15), the patients will be considered for eligibility to receive standard of care. We assume that the decline in HCV viral load would substantially improve the chances of SVR as the reduction of viral load should both increase the efficacy of PR and reduce the odds of drug resistance to HCV-specific protease inhibitor.

* Trial with medicinal product

ELIGIBILITY:
Inclusion criteria:

* Age greater or equal 18 years
* HIV-HCV co-infection
* HCV Genotype 1 infection
* At least one liver biopsy since diagnosis of HCV-infection
* Fibrosis score METAVIR = 2 documented by biopsy OR a stiffness greater or equal 7.0 kPa documented by fibroscan during the previous 12 months.
* Documented previous null-response or partial-response to SOC

Exclusion criteria:

* Contraindications to the study drug under study, e.g. known hypersensitivity or allergy to any ingredient of the study drug
* Patients in need of ART with HIV virological failure (= 400 copies/ml) in the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-04; Primary Completion 2014-04 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Frequency of adverse events during iSIL treatment. | Day 15 (after 14days of treatment)
  The participants will be followed for the duration of study-drug administration and one day follow-up, which counts for 15days
Kinetics of the decline in HCV-RNA after 2 weeks of iSIL treatment (difference in IU/ml from day 1 to day 15). | Day 15
  The participants will be followed for the duration of study-drug administration and one day follow-up, which counts for 15days

SECONDARY OUTCOMES:
Drug levels of iSIL and its influence on the drug-level of co-administrated ART. | Day 15
  The participants will be followed for the duration of study-drug administration and one day follow-up, which counts for 15days
Proportion of patients with HIV virological failure, i.e. confirmed viremia >50cp/ml. | Day 15
  The participants will be followed for the duration of study-drug administration and one day follow-up, which counts for 15days

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Braun, MD, Principal Investigator — University Hospital Zurich, Division of Infectious Diseases and
Locations (1):
- Division of Infectious Diseases and Hospital Epidemiology, University Hospital Zurich, University of Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Braun DL, Rauch A, Aouri M, Durisch N, Eberhard N, Anagnostopoulos A, Ledergerber B, Mullhaupt B, Metzner KJ, Decosterd L, Boni J, Weber R, Fehr J; Swiss HIV Cohort Study. A Lead-In with Silibinin Prior to Triple-Therapy Translates into Favorable Treatment Outcomes in Difficult-To-Treat HIV/Hepatitis C Coinfected Patients. PLoS One. 2015 Jul 15;10(7):e0133028. doi: 10.1371/journal.pone.0133028. eCollection 2015. PMID 26176696